CLINICAL TRIAL: NCT05474079
Title: The Effects of Supervised Exercise Training in the Primary Prevention of Cardiovascular Disease in Stain-Users and Non Statin-Users
Brief Title: Exercise Training & Statins for Cardiovascular Health
Acronym: EXSTATIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiff Metropolitan University (Other)
Collaborators: Health and Care Research Wales (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: STA- 5035
Record Dates: First submitted 2022-03-01; First posted 2022-07-26 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Risk Reduction; Cardiovascular Diseases
MeSH Terms: conditions — Risk Reduction Behavior; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Statin users exercise intervention (Experimental): The exercise training program will consist of individually tailored, progressive moderate-intensity aerobic exercise. Exercise training will comprise of a combination of treadmill, cross-trainer and cycle ergometer-based exercise. Exercise will progressively increase in both intensity and duration throughout the course of the intervention. Participants will begin the intervention with 30 minutes of moderate-intensity aerobic exercise at 40% heart rate reserve (HRR) three times per week for the initial 4 weeks. From week 4, exercise intensity will increase to 50% HRR, and at week 6 the duration of each session will increase to 45 minutes. From week 8, participants will exercise at an intensity of 60% HRR for 45 minutes, and from week 10, this will increase to five sessions per week.
  Interventions: Other: Moderate intensity exercise training
- Statin users conventional care control (No Intervention): Participants randomized to the conventional primary care control group will not receive any supervision or guidance throughout the 12-week intervention beyond the initial standard healthcare advice provided by their general practitioner (GP).
- Non-statin users exercise intervention (Experimental): The exercise training program will consist of individually tailored, progressive moderate-intensity aerobic exercise. Exercise training will comprise of a combination of treadmill, cross-trainer and cycle ergometer-based exercise. Exercise will progressively increase in both intensity and duration throughout the course of the intervention. Participants will begin the intervention with 30 minutes of moderate-intensity aerobic exercise at 40% HRR three times per week for the initial 4 weeks. From week 4, exercise intensity will increase to 50% HRR, and at week 6 the duration of each session will increase to 45 minutes. From week 8, participants will exercise at an intensity of 60% HRR for 45 minutes, and from week 10, this will increase to five sessions per week.
  Interventions: Other: Moderate intensity exercise training
- Non-statin users conventional care control (No Intervention): Participants randomized to the conventional primary care control group will not receive any supervision or guidance throughout the 12-week intervention beyond the initial standard healthcare advice provided by their GP.

INTERVENTIONS:
Other: Moderate intensity exercise training — The exercise training program will consist of individually tailored, progressive moderate-intensity aerobic exercise. Exercise training will comprise of a combination of treadmill, cross-trainer and cycle ergometer-based exercise. Exercise will progressively increase in both intensity and duration throughout the course of the intervention. Participants will begin the intervention with 30 minutes of moderate-intensity aerobic exercise at 40% HRR three times per week for the initial 4 weeks. From week 4, exercise intensity will increase to 50% HRR, and at week 6 the duration of each session will increase to 45 minutes. From week 8, participants will exercise at an intensity of 60% HRR for 45 minutes, and from week 10, this will increase to five sessions per week.
  Arms: Non-statin users exercise intervention; Statin users exercise intervention

SUMMARY:
Cardiovascular disease (CVD) refers to any condition that affects the heart and/or blood vessels (e.g. heart attack, stroke) and is the leading cause of death and disability worldwide. Regular exercise and statin therapy are widely recommended as frontline prevention strategies to reduce CVD risk. Recent changes to National Health Service (NHS) healthcare guidelines state that even individuals with a relatively low risk of CVD (≥10% risk score) should take a statin. When prescribed after a heart attack or stroke, both exercise and statins reduce the risk of a CVD-related death by ~25%, with some evidence to suggest that the combination of these therapies may offer additive cardiovascular protection. However, far less is known about the combined effects of exercise and statin therapy in primary CVD prevention (i.e. before a CVD event). Poor blood vessel function represents the earliest stage of CVD, which can be measured with ultrasound at different regions of the body (limbs, brain, heart) to sensitively detect early CVD risk. Regular exercise provides a variety of cardiovascular benefits and has a direct therapeutic effect on blood vessel function. In contrast, statin therapy primarily reduces CVD risk by lowering cholesterol, which may also improve blood vessel function. Although both therapies can separately reduce CVD risk, the interaction between exercise training and statin therapy on blood vessel function has never been directly compared in the setting of primary prevention, and it's currently unknown whether a combination of both therapies offers additional cardiovascular benefit. Therefore, the main aims of this study are to (i) investigate the effect of supervised exercise training on blood vessel function (limbs, brain, heart) in individuals with a CVD-risk score of ≥10% and (ii) examine whether these exercise effects differ in individuals taking a statin compared to those not taking a statin.

DETAILED DESCRIPTION:
Over 340,000 people in Wales live with cardiovascular disease (CVD). It causes 28% of all annual deaths and costs the Welsh NHS £469 million per year (British Heart Foundation, 2019). Physical inactivity causes a third of all CVD cases and only 53% of Welsh adults currently meet the recommended minimum physical activity guidelines (Statistics for Wales, 2019). Accordingly, Wales is the most physically inactive nation in the UK with one of the highest rates of CVD. Regular exercise is widely recommended by GPs as a frontline prevention strategy to reduce CVD-risk. Similarly, statins are also routinely prescribed as part of primary healthcare across the UK to lower cholesterol levels and reduce CVD-risk. Recent changes to NHS primary healthcare guidelines state that even individuals with a relatively low risk of CVD (10-year CVD-risk score ≥10%; QRISK3) should take a statin. When prescribed after a heart attack or stroke, both exercise and statins reduce the risk of a CVD-related death by ~25%; some evidence suggests that the combination of these therapies may offer additive cardiovascular protection. However, far less is known about the combined effects of exercise and statin therapy in primary CVD prevention.

Sensitive ultrasound techniques can be used to examine vascular, cerebrovascular and cardiac structure and function to provide a comprehensive overview of cardiovascular health. Poor vascular function represents the earliest stage of CVD and is more sensitive at detecting CVD risk than traditional risk factors. Regular exercise provides a variety of cardiovascular benefits and has a direct therapeutic effect on vascular function. In contrast, statin therapy primarily reduces CVD-risk by lowering cholesterol, which may also improve vascular function. Although both therapies can separately reduce CVD risk, the interaction between exercise training and statin therapy on vascular function has never been directly compared in the setting of primary prevention; and it is currently unknown whether a combination of both therapies offers additional cardiovascular benefit.

This study will utilise a comprehensive series of cutting-edge vascular, cerebrovascular and cardiac ultrasound techniques to examine the effectiveness of exercise and statin therapy as primary CVD prevention strategies. If results demonstrate that exercise training provides similar cardiovascular benefits to statin therapy, and/or the combination of these preventive strategies offer additive benefit, this could have considerable implications on primary prevention healthcare recommendations.

ELIGIBILITY:
Inclusion Criteria:

Statin Users:

* Sedentary
* Non-smokers
* 50-65 years old
* A 10-year CVD-risk score > 10% (estimated via QRISK3)
* Weight stable (<5% weight change over the last 3 months)
* Prescription of an 3-hydroxy-3-methylglutaryl coenzyme A reductase (HMG-CoA) inhibitor (statin) in stable dose for a minimum of 3 months and maximum of 3 years

Non-Statin Users:

* Sedentary
* Non-smokers
* 50-65 years old
* A 10-year CVD-risk score > 10% (estimated via QRISK3)
* Weight stable (<5% weight change over the last 3 months)

Exclusion Criteria (Statin Users and Non-Statin Users):

* History or signs/symptoms of established cardiovascular, metabolic, renal or musculoskeletal disease
* Diagnosed with familial hyperlipidaemia and/or diabetes mellitus
* Stage 2 hypertension (≥160/100 mmHg)
* Any contraindications to exercise (e.g. unstable angina, severe orthopaedic conditions) and/or advised by GP not to undertake exercise
* BMI >40kg/m2
* Current smoker or within 6 months of cessation
* Use of any medication other than statins (e.g., fibrates, metformin, thiazolidinediones, orlistat, anti-hypertensives) that could independently alter lipid metabolism and/or vascular function
* Post-menopausal female and using hormone replacement therapy, or pre-menopausal using oral contraceptives that independently alter lipid metabolism and/or vascular function

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-07-20 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in Flow Mediated Dilatation (FMD) | Pre and post intervention (12 weeks)
  Brachial artery FMD, as a non-invasive measure of endothelial nitric oxide function, will be assessed using high resolution Duplex vascular ultrasonography in accordance with published guidelines.

SECONDARY OUTCOMES:
Change in sublingual glyceryl trinitrate (GTN) induced dilatation | Pre and post intervention (12 weeks)
  Sublingual Glyceryl Trinitrate (GTN): Following 10 minutes of supine rest, endothelium independent vasodilator function will be assessed simultaneously in the brachial and carotid artery. A 1-minute baseline recording of the brachial and carotid artery will be acquired on the same high-resolution ultrasound device before sublingual administration of glyceryl trinitrate (GTN; 400µg). GTN is a nitric oxide donor that will cause the arteries to vasodilate allowing a short-lived increase in blood flow. Both the brachial and carotid artery will be imaged for 10-minutes following the administration of GTN and peak diameter and blood flow will be recorded. GTN has been used for many decades in clinical and research work in this and other populations.
Change in cold pressor induced dilatation | Pre and post intervention (12 weeks)
  Cold Pressor Test: Following 15 minutes supine rest, carotid artery reactivity (CAR) to a sympathetic stimulation produced by the cold pressor test (CPT) will be measured. The same ultrasound probe will be repositioned onto the participant's neck and an image of the carotid artery will be recorded continuously for one minute before and then during 3 minutes of hand-to-wrist submersion in ice cold water (4 °C). After the 3 minute CPT, the participant will then remove their hand from the cold water and we will continue to image the carotid artery for an additional 3 minutes. Peak carotid artery diameter and blood flow velocity, and the time taken to reach these peaks during the CPT will be recorded. This procedure has been shown to be reliable and well tolerated in this population.
Change in arterial stiffness | Pre and post intervention (12 weeks)
  Carotid - femoral pulse wave velocity (CF-PWV) will be recorded following 15 minutes of supine rest via applanation tonometry. This measure is the accepted gold standard for non-invasive measurement of arterial stiffness and has been previously validated in this population. The arterial wave form will be recorded at the wrist, neck and groin using a high fidelity micromanometer tipped probe and gated to a 3-lead ECG for measurement of PWV via the SphygmoCor system (SphygmoCor, AtCor-Medical, Sydney, Australia). Pulse wave analysis (PWA) will also be used to measure aortic pressure using the SphygmoCor system.
Change in ultrasound assessment of cerebrovascular function- Assessment of cerebrovascular reactivity | Pre and post intervention (12 weeks)
  Participants will then return to the assessment bed and lay supine for 10 minutes. Following this, participants will perform a carbon dioxide breathing challenge. The protocol will involve the participants breathing a fixed gas mixture of otherwise normal atmospheric air that has a mildly elevated fractional concentration of carbon dioxide (6%). This technique has been routinely used within this population and published guidelines will be followed. Normal atmospheric oxygen content is maintained throughout. Participants will be fitted with a face mask covering their nose and mouth with a one-way valve to prevent rebreathing. An elevation in the fractional concentration of carbon dioxide will be applied for 6 minutes and cerebrovascular blood flow will be measured continuously throughout this protocol, as per published guidelines. This procedure enables the maximal dilation capacity of the cerebrovascular blood vessels to be assessed.
Change in ultrasound assessment of cerebrovascular function -Dynamic cerebral autoregulation | Pre and post intervention (12 weeks)
  Participants will perform a cyclical squat-to-stand protocol. Participants will start in a standing position and then adopt a squat position where the back of their legs are at a ~90◦ angle. This manoeuvre will be repeated and performed at frequency of 10 seconds of squatting, followed by 10 seconds of standing. The duration of the protocol will be 5 minutes. This technique has been used routinely in older populations and is well tolerated and validated.
Change in ultrasound assessment of cerebrovascular function - Cerebrovascular reactivity to an acute bout of exercise | Pre and post intervention (12 weeks)
  After 15 minutes of rest, participants will perform a 10 - 15 minute bout of moderate intensity exercise at 50% predicted heart rate reserve (HRR) on a cycle ergometer.
Change in ultrasound assessment of cerebrovascular function - Assessment of neurovascular coupling | Pre and post intervention (12 weeks)
  Localised changes in cerebrovascular blood flow will be assessed during neuronal activation. The occipital lobe will be activated using a visual stimulus of a flashing checkerboard and participant's will then perform a series of short and repetitive sensory tasks. Sensory stimulation tasks will involve a simple cyclical eye opening and closing protocol, reading a short passage from an non-emotive text book and performing a simple visualisation cognitive task. This technique is frequently used in older populations and a standardised and validated protocol will be adopted.
Change in Cognitive Function Assessment | Pre and post intervention (12 weeks)
  Cognitive Function Assessment: Participants will be asked to complete the Montreal Cognitive Assessment. This paper-based assessment has been validated in this population and examines short term memory, visuospatial abilities, executive functions, attention, concentration and working memory, language and orientation to time and place. The test is scored based on a minimum score of 0 to a maximum score of 30, where a score of >26 is regarded as 'normal cognitive function' and a score of <26 indicative of mild cognitive impairment.
Change in blood lipid profile | Pre and post intervention (12 weeks)
  A 30ml blood sample will be taken from a vein in the arm and analysed for markers of cardiovascular risk. Blood samples will be analysed using the Randox Dayton+ analyser with standard proprietary reagents for total cholesterol, high-density lipoprotein, triglyceride (all lipid measures in mmol). Low-density lipoprotein will then be calculated using according to the Friedwald formula (mmol).
Change in blood glucose and insulin profile | Pre and post intervention (12 weeks)
  A 30ml blood sample will be taken from a vein in the arm and analysed for markers of cardiovascular risk. Blood samples will be analysed using the Randox Dayton+ analyser with standard proprietary reagents for glucose and insulin assayed using commercially available radioimmunoassay (both measures in mmol). Using fasting glucose and insulin concentrations, we then will calculate steady-state beta cell function and insulin resistance via the homeostasis model assessment.
Changes in blood pro-inflammatory cytokines | Pre and post intervention (12 weeks)
  A 30ml blood sample will be taken from a vein in the arm and simultaneously analysed for pro-inflammatory cytokines; Interleukin-1α, Interleukin-1β, Interleukin-6, Interleukin-8, Interleukin-10 Interferon-γ and Tumour Necrosis Factor-α,(all measured in pg/ml) using high sensitivity multiplex enzyme-linked immunosorbent assays (ELISA).

OTHER OUTCOMES:
Change in 7-day physical activity monitoring: Intensity of activity | Pre and post intervention (12 weeks)
  Each participant will be issued with a small lightweight tri-axial accelerometer (activPAL Professional Physical Activity Monitor Technologies Ltd., Glasgow, UK), that will examine 7-day habitual physical activity levels. This device will be worn around the participant's waist continuously for seven consecutive days and will assess and monitor any physical activity and categorise activity bouts into light, moderate and vigorous intensity activity based on metabolic equivalent of task (METS)/hour/day.
Change in 7-day physical activity monitoring: Frequency of activity | Pre and post intervention (12 weeks)
  Each participant will be issued with a small lightweight tri-axial accelerometer (activPAL Professional Physical Activity Monitor Technologies Ltd., Glasgow, UK), that will examine 7-day habitual physical activity levels. This device will be worn around the participant's waist continuously for seven consecutive days and will assess the frequency of any activity bout (bouts/hour/day).
Change in 7-day physical activity monitoring: Duration of activity | Pre and post intervention (12 weeks)
  Each participant will be issued with a small lightweight tri-axial accelerometer (activPAL Professional Physical Activity Monitor Technologies Ltd., Glasgow, UK), that will examine 7-day habitual physical activity levels. This device will be worn around the participant's waist continuously for seven consecutive days and will assess the duration of any activity bout (mins per bout).
Change in 7-day physical activity monitoring: Frequency of sedentary periods | Pre and post intervention (12 weeks)
  Each participant will be issued with a small lightweight tri-axial accelerometer (activPAL Professional Physical Activity Monitor Technologies Ltd., Glasgow, UK), that will examine 7-day habitual physical activity levels. This device will be worn around the participant's waist continuously for seven consecutive days and will assess and monitor the frequency of any sedentary periods (bouts/hour/day)
Change in 7-day physical activity monitoring: Duration of sedentary periods | Pre and post intervention (12 weeks)
  Each participant will be issued with a small lightweight tri-axial accelerometer (activPAL Professional Physical Activity Monitor Technologies Ltd., Glasgow, UK), that will examine 7-day habitual physical activity levels. This device will be worn around the participant's waist continuously for seven consecutive days and will assess and monitor the duration of any sedentary periods (mins per bout)
Change in 24-hour ambulatory blood pressure | Pre and post intervention (12 weeks)
  participant will be issued with a wearable automated blood pressure monitoring device. This validated Mobil-O-Graph system (IEM Germany) will non-invasively measure 24-hour ambulatory blood pressure, aortic pressure and vascular haemodynamics. A small blood pressure cuff will be placed around the upper arm of the participant and connected to a halter monitor for 24 hours. Clear instructions on how to fit and position this device, as well as guidance on how long this device should be worn will be provided by a member of the research team
Change in VO2peak cardiopulmonary max test | Pre and post intervention (12 weeks)
  Participants will be required to complete a maximal exercise test (maximal oxygen consumption [VO2max] test) on a motorised treadmill . Initially, participants will be required to complete a 2 minute slow walking warm-up. The test will then progressively increase in speed and gradient every 2 minutes until the participant is no longer able to continue the exercise (volitional exhaustion). Throughout this procedure each participant will be required to wear a face mask connected to a gas analyser, allowing breath-by-breath oxygen consumption to be continuously measured Upon completion of the test, the gradient and the speed of the treadmill will be reduced and the participants will perform a cool down for 3-5 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Pugh, Principal Investigator — Cardiff Metropolitan University
Locations (1):
- Cardiff Metropolitan University, Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: No